CLINICAL TRIAL: NCT06510972
Title: Non-inferiority of a Strategy of Continuing Oral Intake Compared With Fasting in Patients With Acute Respiratory Failure at Risk of Tracheal Intubation
Brief Title: Non-inferiority of a Strategy of Continuing Oral Intake Compared With Fasting
Acronym: JEUN-TUBE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: DR230315
Record Dates: First submitted 2024-07-09; First posted 2024-07-19 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Patient in Acute Respiratory Failure; Continuation of Oral Intake

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Strategy for continuing to take oral supplements (Experimental): Patients will be able to ingest any type of liquid or solid food orally, at any frequency and in any quantity they wish, according to their tolerance, with paramedical assistance if necessary. The necessary treatments will be administered orally. The patient may benefit from a glucosed intake at the discretion of the practitioner in charge of the patient. The patient will benefit from regular mouth care. Intravenous and oral fluids will be quantified.
  Interventions: Procedure: Strategy for continuing oral intake
- Fasting strategy (Active Comparator): The patient will not be able to ingest liquids or solid foods. The patient will be given glucose or parenteral nutrition at the discretion of the practitioner in charge of the patient. The patient will receive regular mouth care. Oral treatments that are essential and have no parenteral alternative may be administered under paramedical supervision.
  Interventions: Procedure: Fasting strategy

INTERVENTIONS:
Procedure: Strategy for continuing oral intake — Patients will be able to ingest liquids or solid food orally, at any frequency and in any quantity they wish, according to their tolerance, with paramedical assistance if necessary.
  Arms: Strategy for continuing to take oral supplements
Procedure: Fasting strategy — The patient will not be able to ingest liquids or solid food.
  Arms: Fasting strategy

SUMMARY:
Fasting in the intensive care unit is a crucial issue and has been studied in particular in patients on mechanical ventilation or at the time of weaning. To date, there are no data on fasting in patients with acute respiratory failure hospitalised in the intensive care unit but not intubated.

The nutritional attitude to adopt in these patients is not mentioned in the recommendations on nutrition for intensive care patients, even though it has been proven in the literature that this specific category of patients does not achieve the theoretical calorie targets, particularly as a large proportion of these patients are not fed, whether orally (or per os), enteral via a naso- or oro-gastric tube or parenterally. There is therefore a real rationale for trying to maintain a nutritional intake in patients with acute respiratory failure.

One of the fears of the team caring for a patient in acute respiratory failure is the potential occurrence of false routes.

In addition to false routes, orotracheal intubation of patients requiring mechanical ventilation in intensive care presents a risk of inhalation of gastric contents followed by the potential development of pneumonia.

In the clinical setting, inhalation may not be symptomatic, but may progress to severe pneumonia and acute respiratory distress syndrome, pulmonary fibrosis and therefore be life-threatening.

By analogy, in intensive care, patients at risk of intubation are put on a fast as a preventive measure to limit the risk of a false route and the risk of potential inhalation in the event of intubation. This practice, which is very common on admission to intensive care and continuous care units, has not been studied in the literature and is not the subject of recommendations.

Finally, patients hospitalised in intensive care are subject to numerous discomforts.

The hypothesis put forward is that the continuation of intravenous fluids in intensive care units for patients at risk of intubation does not increase the need for intubation and does not increase adverse effects such as false routes or inhalation of gastric contents in patients who ultimately require intubation.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 18 years old
* Participant affiliated to a social security scheme
* Express oral consent of the participant, or failing that of the trusted support person, or failing that of the next of kin
* Patient hospitalised in an intensive care unit or in a continuous surveillance unit or in an intensive care unit for less than 24 hours.
* Criteria for acute hypoxaemic respiratory failure defined as.

  * Respiratory rate > 25 cpm or indifferent if SARS-CoV-2 (Severe acute respiratory syndrome coronavirus 2) infection occurred ≥ 1 time since admission.
  * PaO2/FiO2 < 200 mmHg or equivalent SpO2 (oxygen saturation)/FiO2 (fraction of inspired oxygen) i.e. < 235 (measured under at least 10 L/min high concentration mask)

Exclusion Criteria:

* Patient with criteria for immediate intubation:

  * Persistent or worsening respiratory failure (respiratory rate > 40/min, respiratory failure on physical examination, respiratory acidosis with pH (hydrogen potential ) < 7.25, copious tracheal secretions, hypoxia with SpO2 < 90% despite FiO2 > 80% for more than 5 minutes without technical dysfunction).
  * Major haemodynamic failure (need for increasing vasopressor support with instability and hypoperfusion).
  * Neurological failure (Glasgow score < 8).
  * Cardiac or respiratory arrest
* Chronic lung disease: chronic obstructive pulmonary disease (GOLD grade 3 or 4: Global Initiative for Chronic Obstructive Lung Disease) or other chronic lung disease requiring long-term oxygen or ventilation (this does not include a patient undergoing continuous positive nocturnal pressure for sleep apnoea syndrome).
* Contraindications to oral nutrition: known previous swallowing problems or inability to swallow, digestive sutures, admission for inhalation pneumonia, exclusive parenteral nutrition, etc.
* Patients with a nasogastric or orogastric tube, a jejunostomy or a feeding ileostomy
* Patient already on invasive mechanical ventilation on admission
* Limitation of therapies including a decision not to intubate
* Incapacitated adult (guardianship or curators)
* Pregnant, parturient or breast-feeding women
* Tracheostomised patient
* Patient already included for the first time in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 754 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients intubated or dying without intubation within 96 hours of randomisation | From randomisation to 96 hours

SECONDARY OUTCOMES:
Simple verbal scale between 1 and 4 of sensation of thirst and hunger at D1 after randomisation | At Day 1 after randomisation
Mortality at D28 | At Day 28
Time from randomisation to intubation to Day 28 | From randomisation to day 28
Occurrence of vomiting during intubation | Between the start and end of the intubation procedure
Immediate post-intubation salivary amylase and pepsin rates | Immediate post-intubation
Natraemia rates within 4 days of randomisation | From randomisation to day 4
Occurrence of acute renal failure within 4 days of randomisation | From randomisation to day 4
Occurrence of hypoglycaemia within 4 days of randomisation | From randomisation to day 4
Occurrence of at least one nosocomial pneumonia within 28 days of randomisation | From randomisation to day 28
Occurrence of at least one pneumonia acquired under early mechanical ventilation | From randomisation to day 28

CONTACTS AND LOCATIONS:
Overall Officials: Piotr SZYCHOWIAK, MD, Study Director — University Hospital, Orléans
Locations (11):
- France (11):
  - Intensive care, University Hospital, Blois, Blois
  - Intensive care, Hospital, Bourges, Bourges
  - Intensive care, Hospital, Colombes, Colombes
  - Intensive care, Hospital, Dreux, Dreux
  - Intensive care, Hospital, La Roche sur Yon, La Roche-sur-Yon
  - Intensive care, Hospital, Le MANS, Le Mans
  - Intensive care, Hospital, Lille, Lille
  - Intensive care, Hospital, Morlaix, Morlaix
  - Intensive care, Hospital, Nantes, Nantes
  - Intensive care, University Hospital, Orléans, Orléans
  - Intensive care, University Hospital, Tours, Tours